CLINICAL TRIAL: NCT01208688
Title: FES Therapy:Restoring Voluntary Grasping Function in Chronic SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Rick Hansen Foundation (Other)
Responsible Party: Principal Investigator, Milos Popovic, PhD, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-36; SCISN-2009-36
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FES Therapy (Experimental): FES Therapy
  Interventions: Device: FES Therapy
- Conventional Occupational Therapy (Active Comparator): The conventional therapy represents control activities against which FES therapy will be assessed. Conventional occupational therapy includes : a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach;b)task-specific repetitive functional training;c)strengthening and motor control training using resistance to available arm motion to increase strength; d)stretching exercises;e)electrical stimulation applied primarily for muscle strengthening (this is not FES); and f)activities of daily living including self care where the upper limb was used as an assist if appropriate; and caregiver training. Control and treatment group will have 3 sessions per week (business days only) for 13 to 16 weeks (40 treatment sessions in total). Each session will last 60 minutes.
  Interventions: Other: Conventional Occupational Therapy

INTERVENTIONS:
Device: FES Therapy — Treatment group received functional electrical stimulation and control group received conventional occupational therapy.
  Other Names: Neuroprosthesis
  Arms: FES Therapy
Device: FES Therapy — Subjects will be divided into one of two groups: a) subjects that will be trained with neuroprosthesis for grasping and b) the control group. The control group will be administered standard occupational therapies appropriate for recovery of grasping function in SCI subjects. In group a), neuroprosthesis for grasping will be used to train subjects to reach, grasp and manipulate various objects in the activities of daily living.
  Arms: FES Therapy
Other: Conventional Occupational Therapy — The conventional therapy represents control activities against which FES therapy will be assessed. Conventional occupational therapy includes : a) muscle facilitation exercises emphasizing the neurodevelopmental treatment approach;b)task-specific repetitive functional training;c)strengthening and motor control training using resistance to available arm motion to increase strength; d)stretching exercises;e)electrical stimulation applied primarily for muscle strengthening (this is not FES); and f)activities of daily living including self care where the upper limb was used as an assist if appropriate; and caregiver training. Control and treatment group will have 3 sessions per week (business days only) for 13 to 16 weeks (40 treatment sessions in total). Each session will last 60 minutes.
  Arms: Conventional Occupational Therapy

SUMMARY:
The main objective of this study is to determine the effectiveness of a new treatment regime that uses electrical stimulation for the improvement of hand function in persons with spinal cord injuries (SCI). This treatment has been shown to be useful for stroke patients, and our preliminary work indicates that this may also be the case with SCI patients. Our approach to functional electrical stimulation (FES) represents a departure from the established FES approaches, which involve developing assistive devices for permanent, everyday use. Instead, we use FES as a therapeutic intervention that will help individuals with quadriplegia recover voluntary grasping function. Investigators believe that subjects who undergo FES therapy should be able to grasp objects without stimulation once the treatment program is completed.

DETAILED DESCRIPTION:
The primary objective of the present prospective randomized controlled trial is to investigate if the FES therapy would generate similar level of the improvement in hand function in chronic C4 to C7 incomplete and complete SCI individuals as compared to conventional occupational therapy. For the purpose of this study individuals with chronic SCI are those who sustained injury at least 24 months prior to enrolling in the study. The FES or conventional occupational therapy will be administered thrice-weekly for 13 weeks (i.e., 39 sessions in total) to 60 individuals with SCI. Half of the participants will receive the FES therapy and the other half will receive conventional occupational therapy of equal intensity. The secondary objectives are to evaluate if the improvements in hand function will improve participants' activities of daily living skills and their satisfaction with life.

Background and Significance The sudden onset of a traumatic SCI can result in severe impairments in the motor and/or sensory functions of the body and limbs. A significant part of the expenses incurred after SCI are associated with the need of many individuals with SCI to have a caregiver assist them with various daily tasks such as eating, grooming and ambulation. This dependence,besides being financially strenuous for the patients and their families, frequently precipitates psychological problems such as depression, social withdrawal and inactivity.For persons with quadriplegia, hand function is essential for achieving a high level of independence in their activities of daily living. In a recent survey, it was revealed that the majority of people with quadriplegia rate recovery of hand function as the highest priority.FES is one of the most promising approaches towards improving grasping function in SCI individuals with permanent hand impairment. A neuroprosthesis for grasping is a device that can improve or restore the grasping, holding, and releasing functions in persons with SCI [1]. The neuroprosthesis applies FES to artificially generate a muscle contraction by applying short current pulses to motor nerves innervating muscles. FES can be applied to individuals with SCI to help them restore functions such as walking and grasping by contracting groups of paralyzed muscles in an orchestrated manner.Despite the usefulness of neuroprostheses in improving functionality, SCI consumers, their therapists and psychiatrists remain hesitant to use the technology. For instance, Popovic et al. (not the principal investigator) reported that consumers who retained some dexterity without an FES-assisted system hesitated to use the surface FES device to manipulate small objects, even though they gained significant improvements in function when wearing it. Also, some neuroprostheses such as the Freehand system require invasive procedures for their implementation, which is often unappealing to SCI consumers. These issues with FES, along with the mindset that impairments in functionality are permanent, have led to the design of systems that SCI consumers have little interest in using over long periods of time. Our application of the neuroprosthesis for grasping in this proposal presents a departure from this standard and established approach of FES application. The Compex Motion neuroprosthesis, developed by Drs. Popovic (principal investigator) and Keller1,is a flexible device designed to improve grasping function in both SCI and stroke patients. This multi-channel surface stimulation system for grasping provides both palmar and lateral grasps, and holds a number of advantages over other existing neuroprostheses.Firstly, whereas most other systems were designed and used exclusively as permanent orthotic systems for SCI consumers in order to allow them to grasp, the Compex Motion was designed to help retrain voluntary grasping function. Hence, the device is meant to be used as part of the rehabilitation process towards improving functionality as opposed to merely substituting it. Secondly, the Compex Motion is a surface FES system that does not require implanted systems or possesses features that limit flexibility. These features make it a more suitable option for rehabilitation applications, which typically require portable, flexible, non-invasive, and multi-channel FES systems. Thirdly, although the Compex Motion, Handmaster, and Belgrade Grasping-Reaching System have been used to retrain voluntary grasping function in individuals with stroke, only the Compex Motion has been used for this purpose in individuals with SCI. The advantages of the Compex Motion system over other FES systems is its potential for retraining function in SCI patients and the fact that the system's application does not require the long-term support/commitment of clinical and engineering specialists. Recent innovative advances in FES applications, spearheaded by our team, clearly indicate that the short-term, therapeutic intervention of the neuroprosthesis for grasping can enhance voluntary function in individuals with SCI. These studies also suggest that this novel method of applying FES to augment functional improvement has the potential to improve overall physical and psychological well being of persons with SCI.

ELIGIBILITY:
Inclusion criteria:

* traumatic spinal cord lesion between C4 and C7
* injury at least 24 months prior to enrolling in the study.

Exclusion criteria:

* uncontrolled hypertension
* susceptibility to autonomic dysreflexia
* pressure ulcer
* cardiac pacemaker
* skin rash

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
REL Hand Function Test | 45 min

SECONDARY OUTCOMES:
GRASSPGraded Redefined Assessment of Strength Sensibility and Prehension | 60 min
Functional Independence Measures (FIM) | 35 min
Spinal Cord Independence Measure (SCIM) | 35 min
Client perception of treatment | 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Milos R Popovic, Ph.d, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- See also: Rehabilitation Engineering Laboratory — http://www.toronto-fes.ca